CLINICAL TRIAL: NCT00935415
Title: Time-Effect of Montelukast on Protection Against Exercise-Induced Bronchoconstriction
Brief Title: Time-Effect of Montelukast Protection
Acronym: TEMPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Attilio Boner, Universita di Verona
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PPDD1962
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Exercise-Induced Asthma; Asthma
Keywords: asthma; exercise-induced bronchoconstriction; montelukast; clinical protection; children; time effect
MeSH Terms: conditions — Asthma, Exercise-Induced; Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast (Active Comparator): capsules prepared in blindness
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator): matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast — Montelukast 5 mg
  Other Names: Singulair
  Arms: Montelukast
Drug: Placebo — capsules of matching placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to verify MNT time of onset of protection against EIB in asthmatic children by evaluating different time intervals between dosing and challenge, after a single-dose and after three days of once a day MNT administration.

DETAILED DESCRIPTION:
Within few days after a baseline exercise challenge, children was randomized to a double blind, placebo-controlled, three day doses, crossover study design. In practice each eligible patient was randomized by a computer-generated schedule to receive in sequence double-blind treatments with placebo or MNT (5 mg). Patients in sequence 1 received MNT, then crossed over to matching placebo; vice versa the case was for patients in sequence 2. Placebo and active treatments were separated by a 7-10 day wash-out period. Each child was assigned to one out of seven groups in order to perform the exercise challenge at different time intervals from drug administration which occurred always at 8.00 A.M. On day one the challenge was performed in the different groups 1, 2, 3, 4, 5, 6, and 8 hours after drug administration, respectively. Then treatment was continued as a single day dose for three consecutive days and a third challenge was then performed at the same time of the day.

ELIGIBILITY:
Inclusion Criteria:

* children with exercise-induced asthma

Exclusion Criteria:

* viral infections
* montelukast treatment

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
maximal percentage fall in FEV1 after exercise test from the baseline value | at the first and at the third day of single day drug administration

SECONDARY OUTCOMES:
clinical protection | at the first and at the third day of single day drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Attilio Boner, MD, Principal Investigator — Universita di Verona
Locations (1):
- Pediatric Dept Hospital of Bolzano, Bolzano, Italy